CLINICAL TRIAL: NCT03860870
Title: Detectability of Clenbuterol and Physiological Response in Human Skeletal Muscle
Brief Title: Response to Clenbuterol in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CLEN
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: dried blood spots; skeletal muscle biopsies; muscle strength; muscle signaling

STUDY DESIGN:
Intervention Model Description: Two phases:
  First phase sequential Second phase crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: First phase - open label Second phase - double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clenbuterol (Experimental): Subjects ingest 80 micrograms of clenbuterol tablets
  Interventions: Drug: Clenbuterol Oral Product
- Placebo (Placebo Comparator): Subjects ingest placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clenbuterol Oral Product — Subjects ingest 4x20 microgram clenbuterol tablets
  Arms: Clenbuterol
Drug: Placebo — Subjects ingest placebo tablets
  Arms: Placebo

SUMMARY:
Due to the long half-life (~36 hr) of clenbuterol, detection methods such as dried blood spots (DBS) are a potentially suitable method to easily and non-invasively detect doping misuse of this compound for several days after ingestion. If, and how long, the compound can be detected by DBS has not yet been investigated but is of interest due to its potential in doping-control. The aim is to evaluate whether abuse of clenbuterol can be detected at relevant concentration levels in samples obtained using DBS and to assess the physiological response to clenbuterol in skeletal muscle..

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18-40 years of age
* No known contraindications for anabolic drugs (e.g. cancer)

Exclusion Criteria:

* Abnormal ECG
* Steroid abuse
* Ongoing use of prescription medication
* heavy resistance training more than 2 times weekly
* Disease deemed by the MD to infer a risk to participate in the trial

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Blood clenbuterol concentration | Before (baseline) as well as 3, 8, 24, 72, 168 and 240 hours after administration of clenbuterol
  Concentration of clenbuterol in dried blood spots

SECONDARY OUTCOMES:
Blood clenbuterol concentration | Before (baseline) as well as 3, 8, 24, 72, 168 and 240 hours after administration of study drug
  Concentration of clenbuterol in venous blood
Urine clenbuterol concentration | Before (baseline) as well as 3, 8, 24, 72, 168 and 240 hours after administration of study drug
  Concentration of clenbuterol in urine
Muscle strength | Before (baseline) and 2.5 hours after administration of study drug
  Maximal voluntary isometric contraction in N/m2 of the quadriceps
Muscle signalling | Before (baseline) and 2.5 hours after administration of study drug
  Protein kinase A phosphorylation in vastus lateralis biopsies
Plasma K+ | Before (baseline) as well as 2.5 hours after administration of study drug
  Venous plasma K+ concentration
Muscle mTOR signalling | Before (baseline) as well as 2.5 hours after administration of study drug
  mTOR phosphorylation in vastus lateralis biopsies
Metabolic rate | Before (baseline) as well as 2.5 hours after administration of study drug
  Respriatory exchange ratio of oxygen and CO2
Maximal voluntary strength | Before (baseline) and after two-week treatment of study drug
  Maximal voluntary isometric muscle strength of the quadriceps
Body composition | Before (baseline) and after two-week treatment of study drug
  Lean and fat mass during a DXA-scan
Aerobic capacity | Before (baseline) and after two-week treatment of study drug
  Maximal oxygen uptake during maximal exercise

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided